CLINICAL TRIAL: NCT06238739
Title: Impact of Optimal Temperature Control in Body Contouring Surgery: A Non-Randomized Controlled Clinical Trial
Brief Title: Optimal Temperature Control in Body Contouring Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Total Definer Research Group (Other)
Responsible Party: Principal Investigator, Alfredo Hoyos, Chief of Department of Plastic Surgery, Total Definer Research Group
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NormoT001
Record Dates: First submitted 2023-12-09; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Hypothermia; Postoperative Pain; Postoperative Nausea; Postoperative Complications; Postoperative Shivering; Postoperative Hemorrhage
Keywords: Normothermia; Body contouring; Warming blankets; Safety; High-Definition Liposuction
MeSH Terms: conditions — Hypothermia; Pain, Postoperative; Postoperative Nausea and Vomiting; Postoperative Complications; Postoperative Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Placebo Comparator): Standard measures administered to patients
  Interventions: Other: Control - Standard Strategies for hypothermia prevention
- Group 2 (Experimental): Passive measures
  Interventions: Other: Control - Standard Strategies for hypothermia prevention; Other: Fluid warming before infusion and infiltration
- Group 3 (Experimental): Active measures (Blanketrol)
  Interventions: Other: Control - Standard Strategies for hypothermia prevention; Other: Fluid warming before infusion and infiltration; Device: Thermal convection blanket by water flow (Blanketrol)
- Group 4 (Experimental): Active measures (HotDog)
  Interventions: Other: Control - Standard Strategies for hypothermia prevention; Other: Fluid warming before infusion and infiltration; Device: Conductive fabric electric warming device (HotDog)

INTERVENTIONS:
Other: Control - Standard Strategies for hypothermia prevention — Standard temperature management. Patients underwent one-hour pre- and post-operative warming with hot-air warming blankets at 38°C, without any other preoperative or intraoperative thermal protection measure.
  Other Names: Patient warming with Warm-air blankets
Other: Fluid warming before infusion and infiltration — Passive Measures: Patients underwent one-hour preoperative warming with hot air warming blankets at 38°C (100.4°F), operating room (OR) temperature was maintained at a minimum of 21°C (69.8°F), aseptic/antiseptic solutions along with infiltration fluid were all warmed to 38°C (100.4°F), and surgical fields were kept as dry as possible.
  Other Names: Patient warming with Warm-air Blankets
  Arms: Group 2; Group 3; Group 4
Device: Thermal convection blanket by water flow (Blanketrol) — Blanketrol: Patients underwent continuous intra-operative temperature protection, using a thermal convection blanket by water flow (Blanketrol®) at 40°C (104°F).
  Other Names: Fluid warming before infusion and infiltration; Patient warming with Warm-air Blankets
  Arms: Group 3
Device: Conductive fabric electric warming device (HotDog) — HotDog: Patients underwent permanent intra-operative thermal protection measures with conductive fabric electric warming device (HotDog®) at 40°C (104°F).
  Other Names: Fluid warming before infusion and infiltration; Patient warming with Warm-air Blankets
  Arms: Group 4

SUMMARY:
The goal of this clinical trial is to compare different strategies for normothermia prevention in patients undergoing body contouring and other Aesthetic Plastic Surgery procedures. The main question(s) it aims to answer are:

* Do active measures have an impact on preventing hypothermia in patients undergoing cosmetic procedures?
* Does an active normothermia prevention protocol have any impact in the clinical setting?

Four different protocols will be used for patient peroperative preparation for normothermia.

DETAILED DESCRIPTION:
Participants will receive either of four different protocols for normothermia: Group 1 (Control) involved patients with standard temperature management according to regular institutional protocol, without preoperative or intraoperative thermal protection measures. Group 2 (Passive thermal protection measures) had patients who underwent one-hour preoperative warming with hot air at 38°C (100.4°F), the operating room (OR) temperature was maintained at a minimum of 21°C (69.8°F), aseptic/antiseptic solutions along with infiltration fluid were all warmed to 38°C (100.4°F), and surgical fields were kept as dry as possible. In Group 3 (Active thermal protection measures), patients received the same measures as Group 2, adding continuous intraoperative temperature protection, using a thermal convection blanket by water flow (Blanketrol®) at 40°C (104°F). Group 4 (active thermal protection measures) included patients with the same measures as Group 2, adding permanent intraoperative thermal protection measures with conductive fabric electric warming device (HotDog®) at 40°C (104°F).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing body contouring procedures (liposuction or liposculpture), either individually or combined with a maximum of two other major aesthetic procedures involving face, breast, or dermolipectomy.
* Healthy patients without underlying comorbidities (classified as ASA≤II)

Exclusion Criteria:

* Women with BMI >30 kg/m²
* men with BMI >32 kg/m²
* Patients after massive weight loss
* Smokers

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 197 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Hypothermia prevention | Before induction, Immediately after intubation, at the end of surgery (inside the OR), Upon arrival to the recovery room, before discharge.
  Measure the body temperature throughout the procedure
Pain intensity | Intensity of pain (measured in VAS scale) at the awakening at the recovery room and just before discharge.
  Visual analogue scale rating
Chills | Immediately at awakening at the recovery room.
  Yes or NO
Shivering | Immediately at awakening at the recovery room.
  Yes or NO
Recovery Period | Time interval, measured in minutes and hours, commencing from the patient's admittance into the Post-Anesthesia Care Unit (PACU) until their subsequent discharge.
  Time from Operating Room to discharge from the recovery room.
Analgesic requirements | Number of doses of pain medication required during the patient's recovery period at the PACU, between 1-8 hours after surgery.
  Measure the amount of analgesic required for pain control

SECONDARY OUTCOMES:
Cost-effectiveness of each intervention | Throughout the study completion, about 1 week.
  Analysis of overall costs and effects on patient recovery among the different groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Dhara clinic, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: Yes
Depending upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after publication.
Access Criteria: Request to the main author

REFERENCES:
- [Result] Hoyos AE, Duran H, Cardenas-Camarena L, Bayter JE, Cala L, Perez M, Lopez A, Talleri G, Dominguez-Millan R, Mogollon IR. Use of Tranexamic Acid in Liposculpture: A Double-Blind, Multicenter, Randomized Clinical Trial. Plast Reconstr Surg. 2022 Sep 1;150(3):569-577. doi: 10.1097/PRS.0000000000009434. Epub 2022 Jun 28. PMID 35759637
- [Result] Enrique Bayter-Marin J, Cardenas-Camarena L, Pena WE, Duran H, Ramos-Gallardo G, Robles-Cervantes JA, McCormick-Mendez M, Rocio Gomez-Gonzalez S, Liliana Plata-Rueda E. Patient Blood Management Strategies to Avoid Transfusions in Body Contouring Operations: Controlled Clinical Trial. Plast Reconstr Surg. 2021 Feb 1;147(2):355-363. doi: 10.1097/PRS.0000000000007524. PMID 33565826
- [Result] Bayter-Marin JE, Cardenas-Camarena L, Duran H, Valedon A, Rubio J, Macias AA. Effects of Thermal Protection in Patients Undergoing Body Contouring Procedures: A Controlled Clinical Trial. Aesthet Surg J. 2018 Mar 14;38(4):448-456. doi: 10.1093/asj/sjx155. PMID 29087444